CLINICAL TRIAL: NCT00562640
Title: A Phase I Dose Escalation Safety and Feasibility Study of WT1-Specific T Cells for the Treatment of Patients With Advanced Ovarian, Primary Peritoneal, and Fallopian Tube Carcinomas
Brief Title: Autologous T Cells With or Without Cyclophosphamide and Fludarabine in Treating Patients With Recurrent or Persistent Advanced Ovarian Epithelial Cancer, Primary Peritoneal Cavity Cancer, or Fallopian Tube Cancer (Fludarabine Treatment Closed as of 12/01/2009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 06-155; MSKCC-06155
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2021-08

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent primary peritoneal cavity cancer; stage IIIA primary peritoneal cavity cancer; stage IIIB primary peritoneal cavity cancer; stage IIIC primary peritoneal cavity cancer; stage IV primary peritoneal cavity cancer; recurrent fallopian tube cancer; stage IIIA fallopian tube cancer; stage IIIB fallopian tube cancer; stage IIIC fallopian tube cancer; stage IV fallopian tube cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; 06-155
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Filgrastim; Cyclophosphamide

ARMS (1):
- WT1-Specific T Cells (Experimental): This is a phase I dose escalating trial designed to identify tolerable, clinically active doses of Wilms' tumor gene (WT1) peptide sensitized T cells when administered alone or with nonmyelosuppressive chemotherapy in patients with recurrent or persistent, evaluable WT1+ ovarian, primary peritoneal, or fallopian tube carcinomas.
  Interventions: Biological: filgrastim; Biological: therapeutic autologous lymphocytes; Drug: cyclophosphamide; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: filgrastim — Stem cell mobilization and harvest: Patients receive filgrastim (G-CSF) subcutaneously daily for five days. PBMC are collected by leukapheresis on the fifth day and then cryopreserved for subsequent reinfusion into the patient, in the event of prolonged cytopenia.
Biological: therapeutic autologous lymphocytes — Autologous T-cell infusion with or without conditioning chemotherapy ( fludarabine treatment closed as of 12/01/2009): Approximately 4-6 weeks after T-cell sensitization, patients receive an infusion of autologous WT1-specific T cells over 5-10 minutes on day 0. Patients enrolled in dose levels II and III also undergo pre-infusion lymphodepletive conditioning comprising cyclophosphamide IV on day -2 and fludarabine phosphate IV over approximately 30 minutes on days -6 to -2. After a 48-hour rest period, patients receive autologous WT1-specific T cells. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients with responsive or stable disease after completion of therapy, may receive additional courses of autologous WT1-specific T cells every 14 days.
Drug: cyclophosphamide — Patients enrolled in dose levels II and III also undergo pre-infusion lymphodepletive conditioning comprising cyclophosphamide IV on day -2
Other: laboratory biomarker analysis — Obtained prior to adoptive therapy to quantitate baseline levels of WT1 reactive T cells, by quantitation of WT1 specific CTLp by LDA, T cells secreting IFNγ in response to peptide and, in HLA A0201+ patients, T cell binding WT1 peptide HLA A2 tetramers.
  Other Names: After completion of study therapy, patients are followed for up to 12 weeks.

SUMMARY:
RATIONALE: Giving colony-stimulating factors, such as G-CSF, helps stem cells move from the bone marrow to the blood so they can be collected. Treating stem cells collected from the patient's blood in the laboratory may increase the number of immune cells that can mount an immune response against the tumor. The treated stem cells may help destroy any remaining tumor cells (graft-versus-tumor effect). Chemotherapy may also be given to the patient to prepare the bone marrow for the stem cell transplant.

PURPOSE: This phase I trial is studying the side effects and best dose of autologous T cells when given with or without cyclophosphamide and fludarabine in treating patients with recurrent or persistent advanced ovarian epithelial cancer, primary peritoneal cavity cancer, or fallopian tube cancer. (fludarabine treatment closed as of 12/012009)

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the safety and tolerability of in vitro expanded autologous WT1 specific T cells, when administered alone or in combination with non-myeloablative, immunosuppressive conditioning, in patients with recurrent or persistent, advanced, WT1-positive, ovarian epithelial cancer, primary peritoneal cavity cancer, or fallopian tube cancer.
* To determine the maximum tolerated dose of autologous WT1 specific T cells in these patients.
* To quantitate alterations in the concentration of WT1 specific T cells in the blood at defined intervals post infusion with or without non-myeloablative, immunosuppressive conditioning in order to gain estimates regarding their survival and proliferation.
* To assess the effects of the adoptively transferred T cells on the growth and progression of advanced ovarian epithelial cancer, primary peritoneal cavity cancer, or fallopian tube cancer.

OUTLINE: This is a dose-escalation study of WT1 peptide-specific T cells.

* T-cell generation and isolation: Patients undergo collection of peripheral blood stem cells (PBMC) from which T cells are purified, stimulated in vitro with WT1 peptide-pulsed autologous EBV BLCL, and expanded ex vivo.
* Stem cell mobilization and harvest: Patients receive filgrastim (G-CSF) subcutaneously daily for five days. PBMC are collected by leukapheresis on the fifth day and then cryopreserved for subsequent reinfusion into the patient, in the event of prolonged cytopenia.
* Autologous T-cell infusion with or without conditioning chemotherapy ( fludarabine treatment closed as of 12/01/2009): Approximately 4-6 weeks after T-cell sensitization, patients receive an infusion of autologous WT1-specific T cells over 5-10 minutes on day 0. Patients enrolled in dose levels II and III also undergo pre-infusion lymphodepletive conditioning comprising cyclophosphamide IV on day -2 and fludarabine phosphate IV over approximately 30 minutes on days -6 to -2. After a 48-hour rest period, patients receive autologous WT1-specific T cells. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients with responsive or stable disease after completion of therapy, may receive additional courses of autologous WT1-specific T cells every 14 days.

Blood samples are obtained at baseline and periodically during study and assayed for alterations in circulating levels of WT1 peptide-specific T cells, for biochemical indices of tumor burden, and for radiologic evidence of tumor response. Serum CA125 levels are measured and the number of T cells generating interferon gamma in response to autologous EBV BLCL is quantitated.

After completion of study therapy, patients are followed for up to 12 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed ovarian epithelial carcinoma, primary peritoneal cavity carcinoma, or fallopian tube carcinoma

  * Recurrent or persistent disease after treatment with platinum-based chemotherapy

    * Must have platinum-resistant or intolerant disease
* Evaluable disease, as demonstrated by serological (i.e., CA 125), radiological, or pathological studies
* Tumor must express the Wilms Tumor Gene 1 (WT1) peptide, as detected by IHC analysis of banked (i.e., paraffin-embedded) or freshly biopsied tumor nodules

  * Only WT1 tumors graded as moderate to strong (scores 4-12) according to adapted German Immunoreactive Score criteria are considered positive
* No prior or concurrent brain metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 70-100% OR WHO PS 0-1
* Life expectancy ≥ 6 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60mL/min
* ALT and AST ≤ 2.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* Adequate pulmonary and cardiac function
* No clinical evidence of cardiopulmonary disease, which, in the opinion of the investigator, would preclude enrollment
* Able to keep scheduled visits
* No known hepatitis B or C infection
* No known HIV positivity
* No evidence of bowel obstruction
* No clinically significant heart disease (New York Heart Association class III or IV)
* No active infections requiring antibiotics within two weeks of study entry
* No serious intercurrent illness requiring hospitalization
* No history of primary or secondary immunodeficiency or autoimmune disease
* No other cancers except nonmelanomatous skin cancer within the past 5 years
* Not pregnant or lactating
* No other issue which, in the opinion of the treating physician, would make the patient ineligible for the study

PRIOR CONCURRENT THERAPY:

* More than 3 weeks since prior anticancer therapy (i.e., chemotherapy, biologic therapy, or immunotherapy)
* No history of whole abdominal radiation therapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10-16 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roisin O'Cearbhaill, MB, BCh, Principal Investigator — Memorial Sloan Kettering Cancer Center; Richard J. O'Reilly, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Kyi C, Doubrovina E, Zhou Q, Kravetz S, Iasonos A, Aghajanian C, Sabbatini P, Spriggs D, O'Reilly RJ, O'Cearbhaill RE. Phase I dose escalation safety and feasibility study of autologous WT1-sensitized T cells for the treatment of patients with recurrent ovarian cancer. J Immunother Cancer. 2021 Aug;9(8):e002752. doi: 10.1136/jitc-2021-002752. PMID 34433633
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- WT1 Specific T Cells 5 x 10^6/m2; WT1 Specific T Cells 2 x 10^7/m2; WT1 Specific T Cells 5 x 10^7/m2; WT1 Specific T Cells 1 x 10^8/m2: This is a phase I dose escalating trial designed to identify tolerable, clinically active doses of Wilms' tumor gene (WT1) peptide sensitized T cells when administered alone or with nonmyelosuppressive chemotherapy in patients with recurrent or persistent, evaluable WT1+ ovarian, primary peritoneal, or fallopian tube carcinomas.
Period: Overall Study
Arm/Group | WT1 Specific T Cells 5 x 10^6/m2 | WT1 Specific T Cells 2 x 10^7/m2 | WT1 Specific T Cells 5 x 10^7/m2 | WT1 Specific T Cells 1 x 10^8/m2
Started | 3 | 3 | 4 | 2
Completed | 3 | 2 | 3 | 2
Not Completed | 0 | 1 | 1 | 0
Not completed — Death | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WT1 Specific T Cells 5 x 10^6/m2 | WT1 Specific T Cells 2 x 10^7/m2 | WT1 Specific T Cells 5 x 10^7/m2 | WT1 Specific T Cells 1 x 10^8/m2 | Total
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 12
Age, Continuous [Median (Full Range); unit: years] | 64 [23 to 69] | 52 [47 to 61] | 63.5 [54 to 69] | 63 [54 to 72] | 61 [23 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 2 | 12
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 4 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 4 | 2 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 4 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Assessed for Safety and Tolerability as Assessed by NCI CTCAE v3.0
Description: Participant toxicity will be evaluated by using NCI CTCAE v3.0
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | WT1 Specific T Cells 5 x 10^6/m2 | WT1 Specific T Cells 2 x 10^7/m2 | WT1 Specific T Cells 5 x 10^7/m2 | WT1 Specific T Cells 1 x 10^8/m2
Number analyzed (Participants) | 3 | 3 | 4 | 2
Participants | 3 | 3 | 4 | 2

2. Primary Outcome: Total Number of Dose Limiting Toxicities/DLT's
Time Frame: 2 years
Measure: Number; unit: Dose Limiting Toxicities/DLTs
Arm/Group | WT1 Specific T Cells 5 x 10^6/m2 | WT1 Specific T Cells 2 x 10^7/m2 | WT1 Specific T Cells 5 x 10^7/m2 | WT1 Specific T Cells 1 x 10^8/m2
Number analyzed (Participants) | 3 | 3 | 4 | 2
Dose Limiting Toxicities/DLTs | 0 | 0 | 0 | 0

3. Primary Outcome: Mean Overall Survival
Time Frame: Up to 3 years
Measure: Mean (Full Range); unit: months
Arm/Group | WT1 Specific T Cells 5 x 10^6/m2 | WT1 Specific T Cells 2 x 10^7/m2 | WT1 Specific T Cells 5 x 10^7/m2 | WT1 Specific T Cells 1 x 10^8/m2
Number analyzed (Participants) | 3 | 3 | 4 | 2
months | 11.7 [1.5 to 21.9] | 5.7 [1 to 12] | 22.5 [1 to 32] | 21.4 [20 to 22.8]

4. Primary Outcome: Best Response
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | WT1 Specific T Cells 5 x 10^6/m2 | WT1 Specific T Cells 2 x 10^7/m2 | WT1 Specific T Cells 5 x 10^7/m2 | WT1 Specific T Cells 1 x 10^8/m2
Number analyzed (Participants) | 3 | 3 | 4 | 2
participants
  Stable Disease | 0 | 0 | 1 | 0
  Progressive Disease | 3 | 3 | 3 | 2
  Not Evaluable | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | WT1 Specific T Cells 5 x 10^6/m2 | WT1 Specific T Cells 2 x 10^7/m2 | WT1 Specific T Cells 5 x 10^7/m2 | WT1 Specific T Cells 1 x 10^8/m2
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 2/2
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WT1 Specific T Cells 5 x 10^6/m2 (N=3) | WT1 Specific T Cells 2 x 10^7/m2 (N=3) | WT1 Specific T Cells 5 x 10^7/m2 (N=4) | WT1 Specific T Cells 1 x 10^8/m2 (N=2)
Death not assoc with CTCAE term - Death NOS (General disorders) | 3 | 3 | 4 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 0
Inf norm ANC/gr1/2 neut-Cellulitis(skin) (Infections and infestations) | 1 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Small bowel obstruction - NOS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Inf norm ANC/gr1/2 neut-Pneumonia(lung) (Infections and infestations) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Pulmonary/upper respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | WT1 Specific T Cells 5 x 10^6/m2 (N=3) | WT1 Specific T Cells 2 x 10^7/m2 (N=3) | WT1 Specific T Cells 5 x 10^7/m2 (N=4) | WT1 Specific T Cells 1 x 10^8/m2 (N=2)
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Inf norm ANC/gr1/2 neut-Cellulitis(skin) (Infections and infestations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 3 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Pain - Pelvis (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Small Bowel Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
White blood cell decreased (Investigations) | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT00562640/Prot_SAP_000.pdf